CLINICAL TRIAL: NCT04554901
Title: The Effect of Cocoa on Platelet Function Profiles in Patients With Stable Coronary Artery Disease in Trinidad and Tobago: The ECLAIR Study
Brief Title: The Effect of Cocoa on Platelet Function Profiles in Patients
Acronym: ECLAIR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of The West Indies (Other)
Responsible Party: Principal Investigator, Naveen Seecheran, Principal Investigator, The University of The West Indies
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CREC-SA.0351/05/2020
Record Dates: First submitted 2020-09-13; First posted 2020-09-18 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Platelet Dysfunction
Keywords: Platelet Dysfunction; Cocoa; Polyphenol
MeSH Terms: interventions — Chocolate

STUDY DESIGN:
Intervention Model Description: Blood samples will be collected from participants in 2 separate instances. Initially, a baseline VerifyNow P2Y12 PRU test assay, followed by a subsequent repeat test 2-week after a 2-week, once-daily 70%, 50g cocoa bar manufactured by The UWI Cocoa Research Institute (14 bars).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cocoa (Other): 2-week, once-daily 70%, 50g cocoa bar manufactured by The UWI Cocoa Research Institute (14 bars)
  Interventions: Dietary Supplement: Cocoa

INTERVENTIONS:
Dietary Supplement: Cocoa — 2-week, once-daily 70%, 50g cocoa bar manufactured by The UWI Cocoa Research Institute (14 bars)

SUMMARY:
The effects of chocolate on cardiovascular health are still a matter of debate. It can potentially favor cardiovascular health through the antioxidative effects of cocoa ingredients, such as polyphenols (present in dark but not white chocolate).

DETAILED DESCRIPTION:
Epidemiologic studies have shown inverse associations between dietary polyphenols (present in dark chocolate and cocoa) and mortality from coronary heart disease. However, the basis for this protective association is uncertain. Food polyphenols such as in cocoa reportedly have antioxidant properties and decrease platelet function in vitro. The goal of the present study was to investigate whether the beneficial antioxidant effect of polyphenol-rich cocoa can induce an improvement of endothelial and platelet function in patients with stable coronary artery disease with known platelet hyperreactivity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with stable coronary artery disease.
2. Patients > 18y of age.

Exclusion Criteria:

1. Patients with T2DM.
2. Patients who already ingest any cocoa-based products.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
P2Y12 Reaction Units | 2-weeks
  P2Y12 Reaction Units pre- and post-Cocoa

CONTACTS AND LOCATIONS:
Locations (1):
- The University of the West Indies, Saint Augustine, North, Trinidad and Tobago

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the corresponding author on request.

REFERENCES:
- [Derived] Seecheran NA, Sukha D, Grimaldos K, Grimaldos G, Richard S, Ishmael A, Gomes C, Kampradi L, Seecheran R, Seecheran V, Peram L, Dookeeram D, Giddings S, Sandy S, Ramlackhansingh A, Raza S, Umaharan P, Tello-Montoliu A, Schneider D. Effect of cocoa (Theobroma cacao L.) on platelet function testing profiles in patients with coronary artery disease: ECLAIR pilot study. Open Heart. 2022 Sep;9(2):e002066. doi: 10.1136/openhrt-2022-002066. PMID 36100318